CLINICAL TRIAL: NCT02732457
Title: Allogeneic Hematopoietic Stem Cell Transplantation in HIV-1 Infected Patients
Acronym: HSCT-HIV
Status: Terminated | Type: Observational
Why Stopped: 5 participants recruited in 7 years (no recruitment since 2015). Due to rare patient population and due to ongoing COVID-19 demands on healthcare systems, it was decided by the Protocol Steering Committee to terminate this study.
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: IVPPHSCT01
Record Dates: First submitted 2016-03-23; First posted 2016-04-08 (Estimated); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: HIV-1 Infection
Keywords: HIV; Persistence; Reservoirs; Stem Cell Transplant; Functional Cure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC, BMMC, lymph-node derived cells
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the impact of allogeneic hematopoietic stem cell transplantations (HSCT) in HIV infected patients on the persistence of HIV and the HIV immune response.

DETAILED DESCRIPTION:
1. To assess the impact of HSCT on the immune response to HIV by measuring HIV specific antigens in peripheral blood (via immune assays such as ELISA and Western blot) longitudinally.
2. To measure the decay of persisting HIV by sequencing and quantitating HIV RNA in plasma, and HIV DNA and RNA in peripheral blood cells including CD4+ T cells and CD4+ T cell subsets, as well as in tissue cells derived from fine needle lymph node aspirates, and/or bone marrow aspirates, and/or rectal tissue.
3. To determine the presence of the CCR5 delta 32 allele in the patient prior to and following HSCT which will provide information regarding the presence of this gene in the donor cells.
4. To correlate these findings to the clinical outcome of the individuals enrolled in this study based on their clinical standard of care assessments following HSCT.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, requiring allogeneic, haematopoietic SCT as determined by their treating Physician (Haematologist).
* Over 18 years of age
* Provision of written, informed consent

Exclusion Criteria:

* In the opinion of the investigator that the patient is not able to provide informed consent
* Hb < 9 (g/dL)
* CD4+ T cell count <100 (cells/µl)
* Serious coagulation abnormalities, platelet count < 50.
* Patients currently taking medications that significantly affect the bleeding time (e.g. warfarine, clexane, FXa antagonists)
* History of allergy to local anaesthetics
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HIV infection requiring a HSCT
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Reduction in HIV-1 DNA levels in CD4+ T cells measured by real-time PCR | 3 years
  HIV-1 DNA in CD4+ T cells will be measured by real-time PCR and reported as HIV-1 DNA copies in 10e6 CD4+ T cells

SECONDARY OUTCOMES:
Reduction in HIV-1 Antigens and Antibodies measured by ELISA and Western Blot | 3 years
  HIV-1 antigens and antibodies (Ag/Ab) in peripheral blood will be measured by 4th generation chemiluminescence microparticle immunoassay (CMIA) and by Western blot (WB).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Polizzotto, MD, Principal Investigator — St Vincent's Hospital, Sydney
Locations (1):
- St Vincent's Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided